CLINICAL TRIAL: NCT01835340
Title: Study to Estimate Central Propofol Effect by Measuring Exhaled Propofol Concentrations in Patients
Brief Title: Breath Gas Measurement of Propofol During Anesthesia in Patients With Endourological Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Draeger (Unknown)
Responsible Party: Principal Investigator, Martin Grossherr, PhD, MD, University of Luebeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NCT01835340
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Urological Disease
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- propofol (Experimental): Propofol Patients will receive propofol anesthesia on the study day
  Interventions: Device: Drug: Propofol Anesthesia Patients will undergo propofol anesthesia.

INTERVENTIONS:
Device: Drug: Propofol Anesthesia Patients will undergo propofol anesthesia.

SUMMARY:
Propofol can be measured continuously in breath gas during anesthesia. This study compares propofol concentration in plasma and breath gas and processed electroencephalographic monitoring (bispectral index) under clinical conditions with patients and total intravenous anesthesia. Target controlled infusion technique is used to deliver adequate propofol concentration in plasma.

ELIGIBILITY:
Inclusion Criteria:

• 18 years of age

* Written informed consent
* Ability and willingness to give written informed consent
* American Society of Anesthesiologists (ASA) risk score I-II

Exclusion Criteria:

* Denial of the patient
* Patients ASA physical status III- IV
* Pregnancy
* Volunteers with history of neurological disease or stroke
* Volunteers with a history of recreational drug abuse
* Volunteers with a history of alcohol abuse
* Known drug allergies
* History of adverse events during general anesthesia
* Total intravenous anesthesia not practicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-10; Primary Completion 2017-12-09 (Actual); Study Completion 2017-12-09 (Actual)

PRIMARY OUTCOMES:
Exhaled propofol (parts per billion) | Continuous measurement over 40 min during the induction of anesthesia and 30 min during recovery of anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Gehring, Professor, Principal Investigator — University of Luebeck
Locations (1):
- Dept. of Anesthesiology and Intensive Care, Lübeck, Schleswig-Holstein, Germany

REFERENCES:
- [Background] Grossherr M, Hengstenberg A, Meier T, Dibbelt L, Igl BW, Ziegler A, Schmucker P, Gehring H. Propofol concentration in exhaled air and arterial plasma in mechanically ventilated patients undergoing cardiac surgery. Br J Anaesth. 2009 May;102(5):608-13. doi: 10.1093/bja/aep053. Epub 2009 Mar 31. PMID 19336539